CLINICAL TRIAL: NCT02696811
Title: Randomised 6-week, Parallel Group, Placebo Controlled Intervention Trial to Investigate the Effects of White Carrots on Inflammatory Markers and Lymphocyte DNA Damage
Brief Title: The Effects of Foods on Cell Damage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VEG_01
Record Dates: First submitted 2016-02-17; First posted 2016-03-02 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2016-02

CONDITIONS: DNA Damage; Inflammation
Keywords: cancer; inflammation; dietary intervention trial
MeSH Terms: conditions — Inflammation; Neoplasms | interventions — falcarinol; falcarindiol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oat biscuits (Placebo Comparator): Participants will eat 3 oat biscuits per day for 6 weeks
  Interventions: Dietary Supplement: Oat biscuits
- White Carrots (Experimental): Participants will eat 100g (cooked weight) of white carrots per day for 6 weeks
  Interventions: Dietary Supplement: White carrots

INTERVENTIONS:
Dietary Supplement: White carrots — White carrots contain compounds called polyacetylenes, including falcarinol, falcarindiol and falcarindiol-3-acetate.
  Other Names: Falcarinol; falcarindiol; falcarindiol-3-acetate
  Arms: White Carrots
Dietary Supplement: Oat biscuits — The 3 oat biscuits contain the same amount of fibre and sugar as the white carrot but without the polyacetylenes.
  Arms: Oat biscuits

SUMMARY:
Studies have shown that certain compounds inside vegetables can reduce the risk of cancer. Carrots in particular have an association with reduced incidence of colorectal, bladder and breast cancer. Compounds in carrots, called polyacetylenes, have been studied in isolated cells that have shown a reduction in cancer cells as well as inflammatory markers which have been associated with an increased risk of cancer. These polyacetylenes have not been well studied in the human body and it is unclear whether they are able to affect the biomarkers of health (disease) including DNA damage and inflammatory markers. The aim of this research project is to determine whether eating a portion of white carrots every day for 6 weeks can lead to a reduction in DNA damage and inflammatory markers compared to a control period of 6 weeks consuming a polyacetylene-free diet and a control food of a high fibre oat biscuit.

ELIGIBILITY:
Inclusion Criteria:

* Non -smokers
* BMI between 18.5 and 30

Exclusion Criteria:

* smoking
* taking anti-inflammatories
* taking aspirin or aspirin-like drugs
* antibiotic use in the last 3 months
* metabolic conditions or conditions affecting the metabolism or digestion

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in lymphocyte DNA damage from baseline after 6 weeks of carrot or oat supplementation in the diet, and after 6 weeks wash out (no carrots or oats). | Baseline measures then 2 periods of 6 weeks (baseline, intervention and wash out)
  Lymphocyte DNA damage will be measured by comet assay. Comet 'tail length' represents the number of single strand breaks in the DNA that leave the nucleus when the cells undergo electrophoresis - the longer the 'tail' the more strand breaks. Tail length will be measured from lymphocyte DNA samples at baseline, after 6 weeks of the intervention period and again after 6 weeks of the wash out period. Statistical analysis will compare the extent of damage after supplementation of carrots or oats in the diet (intervention period) to damage at baseline and to damage after the wash out period.
Change in inflammation from baseline after 6 weeks of carrot or oat supplementation in the diet, and after 6 weeks wash out. | Baseline measures then 2 periods of 6 weeks (baseline, intervention and wash out)
  Inflammatory markers (blood CRP, TNF-alpha, IL-6 and urine PE2M) will be measured by ELISA assay. at baseline, after 6 weeks of the intervention period and again after 6 weeks of the wash out period. Statistical analysis will compare the inflammation levels after supplementation of carrots or oats in the diet (intervention period) to inflammation at baseline and inflammation after the wash out period.

SECONDARY OUTCOMES:
Analysis of faecal water from baseline after 6 weeks of carrot or oat supplementation in the diet, and after 6 weeks wash out to determine toxicity to colon epithelial cells. | Baseline measures then 2 periods of 6 weeks (baseline, intervention and wash out)
  Faecal samples will be collected at baseline, after intervention and after wash-out. Faecal water will be removed from the samples and used in cell culture with colon epithelial cells. After culture, the cells will undergo comet assay to determine the amount of strand breaks that occur in each of the three treatments. Tail length will be measured from colon epithelial cell DNA samples from baseline, intervention period and the wash out period samples. Statistical analysis will compare the extent of damage to epithelial cells after exposure to faecal water made during supplementation of carrots or oats in the diet (intervention period) to damage with baseline and wash out period faecal water.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Brandt, Principal Investigator — Newcastle University
Locations (1):
- Agriculture Building, Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided